CLINICAL TRIAL: NCT05096026
Title: Effect of Electronic and Mail Outreach From Primary Care Physicians for COVID-19 Vaccination Among Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RDO KPNC 21-044
Record Dates: First submitted 2021-10-25; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Vaccination

STUDY DESIGN:
Masking Description: Telephone interviewers were blind to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard PCP Outreach (Experimental): These patients were sent standard outreach messages to promote COVID-19 vaccination.
  Interventions: Behavioral: Standard PCP Outreach
- Culturally Tailored PCP Outreach (Experimental): These patients were sent messages similar to those in the Standard PCP Outreach Group, but with additional culturally tailored content.
  Interventions: Behavioral: Culturally Tailored PCP Outreach
- Usual Care (No Intervention): These patients were not sent the above study outreach messages, but may have received other messages from their local medical centers or counties.

INTERVENTIONS:
Behavioral: Standard PCP Outreach — These patients were sent two study outreach messages. Study Outreach 1 was an electronic secure message sent on behalf of the PCP, encouraging COVID-19 vaccination and designed based on behavioral science principles. Letters were sent to patients who had not signed up for the electronic health record portal. Study Outreach 2 was a postcard sent to all patients who had not been vaccinated or made an appointment by four weeks after Study Outreach 1.
  Arms: Standard PCP Outreach
Behavioral: Culturally Tailored PCP Outreach — These patients were sent messages similar to those in Standard PCP Outreach, but with additional culturally tailored content and photos.
  Arms: Culturally Tailored PCP Outreach

SUMMARY:
This randomized controlled trial tested the effect of culturally tailored and standard electronic secure messages and mailings from patients' primary care physicians to encourage COVID-19 vaccination among adults aged 65 and older.

DETAILED DESCRIPTION:
This randomized controlled trial tested the effect of culturally tailored and standard electronic secure messages and mailings from patients' primary care physicians to encourage COVID-19 vaccination among adults aged 65 and older. Patients who had not received a COVID-19 vaccination or appointment after previous outreach attempts were randomized to receive (a) an electronic secure message and/or mail outreach from their PCP, (b) similar outreach with additional culturally tailored content, or (c) usual care. The primary outcome was receipt of COVID-19 vaccination during the 8 weeks after the initial study outreach date.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Received COVID-19 vaccine prior to Study Outreach 1.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8287 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Days to COVID-19 vaccination | During the 8 weeks after Study Outreach 1 was sent
  Days to COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Lieu, MD, Principal Investigator — The Permanente Medical Group
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on submission of a protocol approved by the Kaiser Permanente Northern California Institutional Review Board or Research Determination Official, and contingent on appropriate data sharing agreement being completed.
Supporting Information: Study Protocol
Time Frame: December 1, 2022 through December 1, 2024
Access Criteria: Deidentified data will be shared on submission of a protocol approved by the Kaiser Permanente Northern California Institutional Review Board or Research Determination Official, and contingent on appropriate data sharing agreement being completed.

REFERENCES:
- [Derived] Lieu TA, Elkin EP, Escobar PR, Finn L, Klein NP, Durojaiye C, Prausnitz S, Quesenberry CP, Sawyer D, Teran S, Goler N, Parodi SM, Chen YI. Effect of Electronic and Mail Outreach From Primary Care Physicians for COVID-19 Vaccination of Black and Latino Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2217004. doi: 10.1001/jamanetworkopen.2022.17004. PMID 35713906